CLINICAL TRIAL: NCT06907992
Title: Short-Course Antifungal Therapy vs Standard of Care (14 Day Therapy) for Uncomplicated Candidemia (SCAT)
Brief Title: A Study Comparing Short-course Antifungal Therapy (SCAT) 7 Day vs Standard 14 Day Antifungal Therapy for Uncomplicated Candidemia
Acronym: SCAT
Status: Not yet recruiting | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Jose Vazquez, Principal Investigator, Augusta University
Other Study IDs: MSG 23; U01CK000692 (NIH)
Record Dates: First submitted 2025-03-25; First posted 2025-04-03 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Candidemia
Keywords: candidemia; uncomplicated candidemia; antifungal therapy; echinocandin; caspofungin; micafungin; rezafungin; anidulafungin
MeSH Terms: conditions — Candidemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 7 Days: Study participants randomized to the 7 Day group will receive the short-course antifungal therapy for 7 days.
  Interventions: Drug: Antifungal treatment
- 14 Days: Study participants randomized to the 14 Day group will receive the standard of care antifungal therapy for 14 days.
  Interventions: Drug: Antifungal treatment

INTERVENTIONS:
Drug: Antifungal treatment — Short-course antifungal therapy (7 days) versus standard of care antifungal therapy (14 days)

SUMMARY:
The goal of this clinical trial is to assess whether a seven-day course of standard of care (echinocandin) antifungal therapy is non-inferior to a 14-day course of echinocandin antifungal therapy in patients with uncomplicated candidemia in terms of clinical, mycologic, adverse events and all cause mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years of age
2. Uncomplicated candidemia (positive blood culture only). No evidence of invasive candidiasis at day 1 or until day 7.
3. Received < 5 days of prior antifungal therapy
4. Informed Consent for randomization
5. Patients that did not consent to randomization have consented to be used as a natural history (controls) and will allow collection of available data from the medical record.

Exclusion Criteria:

1. Inadequate source control (e.g., unable to remove endovascular devices, urinary catheters).
2. Invasive candidiasis of any type (e.g., deep seated candidiasis from sources other than blood)
3. Abnormal LFTs > 10-fold
4. Greater than 5 days of prior antifungal therapy
5. Endovascular devices that cannot be removed.
6. Immunocompromised patients (AIDS/HIV; solid organ transplant, bone marrow transplant patients, oncology patients receiving chemotherapy, neutropenic patients (ANC of < 1,500 cells/L
7. Neutropenic at time of consent (what does this mean)
8. Break-through candidemia (people with prior candidemia who relapsed) after treatment with antifungal therapy)
9. Unable to provide informed consent from either the patient or legally authorized authority (LAR)
10. Expected mortality within 96 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from:
  A. Inpatient settings based on positive blood cultures for candidemia. B. Daily review of microbiology labs C. Referrals from investigators, ICUs and hospital unit personnel
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication of candida from the blood at day 7 or day 14 | 14 Days
  Blood culture monitoring at day 7 and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Jose Vazquez, MD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No